CLINICAL TRIAL: NCT00879099
Title: The Effect of Paroxetine on the Plasma Levels of Timolol Using Ophthalmic 0.5% Timolol Eye Drops and 0.1% Timolol Eye Gel in Healthy Volunteers
Brief Title: Interaction Study of Timolol Eye Drops and Paroxetine Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santen Oy (Industry)
Responsible Party: Auli Ropo, Study director
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 73654; Eudra CT 2008-007324-26
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Interaction; healthy volunteers; Interaction study for healthy volunteers
MeSH Terms: interventions — Paroxetine; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Paroxetine (Active Comparator)
  Interventions: Drug: Paroxetine
- Gelatine capsule (Placebo Comparator)
  Interventions: Drug: Placebo
- Timolol 0.5 % eye drops (Experimental): The plasm levels of timolol will be measured after one drop of timolol has been administered into both eyes.
  Interventions: Drug: timolol maleate
- Timosan 0.1% eye gel (Experimental): The plasm levels of timolol will be measured after one drop of timolol has been administered into both eyes.
  Interventions: Drug: timolol maleate

INTERVENTIONS:
Drug: Paroxetine — Paroxetine 20 mg once a day during two treatment periods. One treatment period lasts for 3 days.
  Arms: Paroxetine
Drug: Placebo — Gelatine capsule once a day during two treatment periods. One treatment period lasts for 3 days.
  Arms: Gelatine capsule
Drug: timolol maleate — Oftan Timolol 0,5 % eye drop. One drop into both eyes on day 3 after taking paroxetine or placebo capsules for three days.
  Arms: Timolol 0.5 % eye drops
Drug: timolol maleate — Timosan 0,1 % eye gel. One drop into both eyes on day 3 after taking paroxetine or placebo capsules for three days.
  Arms: Timosan 0.1% eye gel

SUMMARY:
The aim of the study is to investigate the effect of antidepressant paroxetine, on the plasma levels of timolol and its main metabolites after topical application of ophthalmic timolol products.

This will be a phase I, randomised, 4-phase cross-over study in healthy volunteers. Healthy male volunteers aged 18 - 40 years will be enrolled.

Placebo or paroxetine will be given for three days after which 1 drop of timolol product will be administered once in both eyes.

The duration of the paroxetine or placebo treatment period will be 3 days. There will be four different treatment periods. A washout between the study periods will be at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18 - 40 years of age
* be in good general health
* be willing to follow instructions
* provide a written informed consent
* have a BMI of 18.5 - 26
* have systolic blood pressure at least 105 mmHg
* have haemoglobin at least 135 g/l.

Exclusion Criteria:

* known hypersensitivity to timolol, paroxetine or any component of the study medications
* any contraindications to timolol treatment including asthma and obstructive lung disease
* any contraindications to paroxetine treatment
* have heart rate 50/min or less in rest
* any regular medication
* allergy requiring antihistamine or ocular or nasal treatment
* clinically significant abnormalities (from normal limits) in laboratory values: basic blood count, creatinine, ALAT, AFOS, gamma-GT, K, Na
* clinically significant EKG abnormalities assessed by the investigator
* blood donation within the last 60 days (the required time period between two donations for men given by RedCross Finland).
* participation in another clinical trial involving an investigational drug/device, or participation in such trial within the last 60 days

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary parameters will be timolol area under the plasma drug concentration-time curve (AUC0-12h) and highest drug concentration observed in plasma (Cmax). | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Janne Backman, MD, PhD, Principal Investigator — Department of Clinica Pharmacology, Institute of Clinical Medicine, University of Helsinki
Locations (1):
- University of Helsinki, Department of Clinical Pharmacology, Helsinki, Biomedicum, Finland